CLINICAL TRIAL: NCT05003141
Title: A Phase 1a/1b Study of PSB202 in Patients With Previously Treated-, Relapsed-, Indolent B-Cell Malignancies
Brief Title: PSB202 in Patients With Previously Treated-, Relapsed-, Indolent B-Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Puget Sound Biotherapeutics (dba Sound Biologics) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSB202-01
Record Dates: First submitted 2021-07-20; First posted 2021-08-12 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Follicular Lymphoma; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Waldenstrom Macroglobulinemia; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Indolent Lymphoma; Refractory B-Cell Lymphoma; MALT Lymphoma
Keywords: Phase 1; CD20+; CD37+; B-cell malignancy; B-cell lymphoma; monoclonal antibody
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: Phase 1a: 3+3 dose escalation design Phase 1b: 3 Expansion cohorts (N=20 each). Expansion beyond N=20 in a cohort is predicated on an ORR of at least 35% (Futility threshold) observed in the initial N=20 in the cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-arm, escalating dose levels (Experimental): 3 + 3 Phase 1 dose escalation design; sequential ascending dose levels.
  Interventions: Drug: PSB202

INTERVENTIONS:
Drug: PSB202 — PSB202 is an antibody combination product comprised of two full-length monoclonal antibodies, PSB102 and PSB 107, respectively targeting CD20 and CD37. PSB202 is manufactured to work as a single product.

SUMMARY:
Product: PSB202 is a novel biological entity consisting of two engineered monoclonal antibodies, an Fc-enhanced humanized type II anti-CD20 IgG1 (PSB102) and a humanized anti-CD37 IgG1 (PSB107), that target B-cells. PSB202 is manufactured to work as a single product with the two components of PSB202 enabling a distinct dual target-specific antibody directed cell killing of B-cells.

Study: Multi-center-, International Phase 1a/1b (Escalation/Expansion) study in patients with indolent-, relapsed-, B-cell malignancies. The Phase 1a (Dose Escalation) part of study follows a 3+3 design.

DETAILED DESCRIPTION:
Product: PSB202 is a novel biological entity consisting of two engineered monoclonal antibodies, an Fc-enhanced humanized type II anti-CD20 IgG1 (PSB102) and a humanized anti-CD37 IgG1 (PSB107), that target B-cells. PSB202 is manufactured to work as a single product with the two components of PSB202 enabling a distinct dual target-specific antibody directed cell killing of B-cells.

Study: Multi-center-, International Phase 1a/1b (Escalation/Expansion) study in patients with indolent-, relapsed-, CD20+ and CD37+ expressing B-cell malignancies. Phase 1a (Dose Escalation) portion of study follows 3+3 design. Phase 1b (Expansion) enrolls with up to 20 patients in each one of 3 disease-specific cohorts: (1) FL; (2) CLL/SLL, and (3) a mixed indolent B-cell histology cohort comprising WM, indolent phenotype MCL, and MZL.

Primary objectives for Phase 1a are Safety (DLT) and establishing a recommended Phase 1b dose. Primary objective for Phase 1b is establishing preliminary evidence of an anti-lymphoma response in each of the 3 Expansion cohorts, as determined by ORR.

ELIGIBILITY:
Inclusion Criteria:

Phase 1a (dose escalation):

1. Histologically confirmed CD20+ expressing indolent NHL (defined below), CLL or WM, failed or intolerant to standard of care therapies;
2. Relapsed/refractory following at least 2 prior lines of standard of care treatment. Prior treatments received must be documented on the enrollment request form. For FL, prior treatment must have included at least 1 rituximab containing regimen.
3. First three dose levels: in the opinion of the investigator, able to tolerate potentially subtherapeutic doses of PSB202 for the duration of a 28-day DLT observation window.

   Phase 1b - Dose Expansion:
4. Histologically confirmed CD20+ expression. For CD37+, if unavailable from the chart at screening, CD37+ expression may be documented from a new or archived blood specimen after enrollment.
5. Relapsed indolent NHL: histologies that may be included are CLL/SLL, MZL, MALT-lymphoma, follicular NHL, MCL or WM failed, relapsed/refractory or intolerant to at least 2 standard of care therapies. (APPENDIX B). For FL, prior treatment must have included rituximab. MCL must have received a prior alkylating agent.
6. Patients must have documented disease progression after at least two prior standard-of-care regimens.
7. Patients must have measurable disease.

   All Patients:
8. Signed Informed Consent;
9. Eastern Cooperative Oncology Group (ECOG) 0-2
10. Last dose of any anti-CD20 antibody therapy must have been >4 weeks before the first dose of PSB202
11. Patients with a medical history of Covid-19 positivity at within 6 months prior to enrollment, must be retested within 7 days of enrollment and confirm Covid-19 negativity by a PCR-test.
12. At least 18 years of age. There is no upper age restriction.
13. Four weeks wash-out from any other prior cancer therapy, including rituximab or BTK-inhibitors. However, some heavily pretreated patients are at risk for significant morbidity from accelerated disease progression or "flare" when treatment is discontinued prior to the initiation of subsequent effective therapy. Absent residual toxicity and with documented Medical Monitor approval, such patients may receive study drug after five drug half-lives have passed following discontinuation of the immediate pre-study therapy.
14. Adequate hematologic and coagulation status, defined as the following on C1D1 before treatment:

    1. Absolute neutrophil count (ANC) ≥ 0.75 billion/L; not requiring growth factors; after the DLT period, growth factor support is allowed and considered supportive care.
    2. Platelet count ≥75 billion/L not requiring transfusion support; if there is documented bone marrow involvement, platelet transfusions may be used up to 7 days prior to C1D1 to achieve this threshold.
    3. Hemoglobin (Hb) ≥9 mg/dL not requiring transfusion support or growth factors. After the DLT period, growth factor support is allowed and considered supportive care.
    4. Adequate coagulation, defined as aPTT and PT (INR) not greater than 1.5 × upper limit of normal (ULN) (patients appropriately anticoagulated for a preexisting medical condition [e.g., atrial fibrillation] may be eligible with documented Sponsor approval).
15. Adequate hepatic function, defined as:

    1. ALT or AST ≤2.5 X the ULN or ≤5 X ULN with documented liver involvement.
    2. Total bilirubin ≤1.5 X ULN or ≤3 X ULN with documented liver involvement and/or Gilbert's Disease
    3. Adequate renal function, with estimated glomerular filtration rate (eGFR) ≥50 mL/minute.
16. Ability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation.
17. Willingness of men and women of reproductive potential to observe conventional and effective birth control for the duration of treatment and for 3 months following the last dose of study treatment; this may include barrier methods such as condom or diaphragm with spermicidal gel.

    Exclusion Criteria

    Phase 1a (dose escalation) only:
18. NHL with bulky disease defined as a mass ≥10 cm in longest diameter
19. Transformation (e.g., Richter's transformation, prolymphocytic leukemia, transformed NHL, blastoid lymphoma) prior to planned start of PSB202. In addition, no concurrent investigational therapy is permitted.

    All patients: Phase 1a (dose escalation) and Phase 1b (dose expansion):
20. Major surgery within 4 weeks prior to planned start of PSB202
21. Radiotherapy with a limited field of radiation for palliation within 7 days of the first dose of study treatment, except for patients receiving radiation to more than 30% of the bone marrow or receiving whole brain radiotherapy, which must be completed at least 4 weeks prior to the first dose of study treatment
22. Continuation of certain standard of care anticancer therapies, including hormonal therapy for breast and prostate cancer, and growth factor support after completion of the DLT-period, is allowed.
23. Therapeutic monoclonal antibody treatment must be discontinued a minimum of 4 weeks prior to the first dose of PSB202. PSB202 may be started sooner after prior investigational agent or anticancer therapy if considered by the Investigator to be safe and within the best interest of the patient (e.g., to avoid disease flare) and with documented Sponsor approval.
24. Any unresolved toxicities from prior therapy greater than CTCAE (version 5.0) Grade 2 or greater at the time of starting study treatment except for alopecia.
25. History of autologous stem cell transplant (auto-SCT) or chimeric antigen receptor-modified T cell (CAR-T) therapy within the past 180 days with any of the following: cytopenias from incomplete blood cell count recovery post-transplant, need for anti-cytokine therapy, residual symptoms of neurotoxicity > Grade 1, or ongoing immunosuppressive therapy.
26. Active graft versus host disease (GVHD, including resultant from any prior solid organ transplants, if received), or ongoing immunosuppressive therapy.
27. History of allogeneic stem cell transplant (allo-SCT) or allogeneic CAR-T at any time in the patient's medical history
28. Known central nervous system (CNS) involvement by lymphoma. Patients with previous treatment for CNS involvement who are neurologically stable and without evidence of active CNS-disease may be eligible if a clinical rationale is provided by the Investigator and with documented Sponsor approval
29. Active auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP])
30. Cerebrovascular accident (CVA), Transient ischemic attack (TIA), myocardial infarction, unstable angina, or New York Heart Association (NYHA) class III or IV heart failure < 6 months of study screening; mean ECG QT-interval corrected according to Fridericia's formula (QTcF) > 450 milliseconds (ms) (males) or > 470 ms (females) obtained from three ECGs; uncontrolled arrhythmia < 3 months of study screening. Patients with rate-controlled arrhythmias may be eligible for study entry at discretion of the Investigator.
31. Active uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the Investigator and the Sponsor makes it undesirable for the patient to participate in the trial. Screening for chronic conditions is not required.
32. Tested positive for Human Immunodeficiency Virus (HIV) is excluded (due to potential drug-drug interactions between anti-retroviral medications and PSB202 and risk of opportunistic infections). For patients with unknown HIV status, HIV testing will be performed at Screening
33. Active viral hepatitis (B or C, HBsAg, anti-HBs/HBcAb and anti-HCV Ab tests) as demonstrated by positive serology or requiring treatment. Subjects who are anti-HBs/HBcAb (+) without detectable HBV-DNA are eligible. Subjects with a history of Hepatitis C and have received successful curative treatment are eligible.
34. Pregnancy or lactation.
35. Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
36. History of drug-induced liver injury or cirrhosis
37. History of pneumonitis or interstitial lung disease
38. Patients with significant medical diseases or conditions, as assessed by the Investigator and Sponsor, that would substantially increase the risk-benefit ratio of participating in the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Through study completion; up to 27 weeks
  Adverse Events, defined and graded per NCI Common Toxicity criteria (V5)
Dose Limiting Toxicity (DLT) | 3 weeks
  Defined Grade 3, Grade 4, and Grade 5 events occurring during the DLT-observation period

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 2 months
  Cmax for each of the two antibody components of PSB202 (PSB102 and PSB107)
Area under the Plasma Concentration versus Time Curve (AUC) | 2 months
  AUC for each of the two antibody components of PSB202 (PSB102 and PSB107)
Number of Patients with measurable Anti-Lymphoma Response | Up to 27 weeks
  International Working Group Criteria (Lugano) for NHL; Hallek Criteria for CLL
Change in CD20+ cell counts | 2 months
  Surrogate Pharmacodynamic marker: Change in CD20+ cell counts by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey E. Roeker, MD, Study Chair — Memorial Sloan-Kettering Cancer Center, New York, NY
Locations (5):
- United States (2):
  - Norton Cancer Institute, Louisville, Kentucky
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Australia (2):
  - Epworth Healthcare, East Melbourne, Victoria
  - One Clinical research, Perth, Western Australia
- Ruijin Hospital, Shanghai, China